CLINICAL TRIAL: NCT06059079
Title: Using Higher Cut-off Values to Diagnose Acute Myocardial Infarction in Patients With Elevated Hs-cTnT Concentrations
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Director of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 023
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; High sensitivity cardiac troponin T; Rule in

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elevated hs-cTnT group
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
High-sensitive cardiac troponin T (hs-cTnT) is a cornerstone for diagnosing acute myocardial infarction (AMI). However, it is often challenging to diagnose AMI in patients with elevated hs-cTnT before a rise or fall of hs-cTnT can be observed. The elevations of hs-cTnT are caused not only by AMI, but also by other cardiac or even non-cardiac diseases. Thresholds above the 99th percentile have been proposed to improve the specificity and to accelerate the rule in of myocardial infarction. This study aimed to find a more accurate cut-off value to rule in AMI in patients with elevated hs-cTnT.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is a major cause of morbidity and mortality worldwide. In real clinical practice, early and accurate recognition of AMI is crucial to accelerate effective reperfusion therapy. High-sensitivity cardiac troponin T (hs-cTnT) is an important protein that regulates cardiomyocytes excitability, which can be proliferated in cardiomyocytes and released into the blood after myocardial injury or infarction. According to the fourth universal definition of AMI, a rise and/or fall of cTn values with at least one value above the 99th percentile URL is the essential precondition for diagnosing AMI. However, it is challenging for clinicians to diagnose AMI in patients with elevated hs-cTnT levels before a rise and/or fall of hs-cTnT values can be observed, particularly for those who present atypical symptoms and non-significant changes in electrocardiograms (ECG). When the 99th percentile upper reference limit (URL) is referred, it happens frequently that the elevations of hs-cTnT are not caused by AMI, but by other cardiac or even non-cardiac diseases. Therefore, thresholds above the 99th percentile have been proposed to improve the specificity and to accelerate the rule in of myocardial infarction.

This study aimed to find a higher and more accurate cut-off value of hs-cTnT to rule in AMI in a large volume of patients with elevated hs-cTnT.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized from January 1,2015 to May 31,2023 in the First Affiliated Hospital of Nanjing Medical University with hs-cTnT concentrations over 14.0 ng/L were enrolled.

Exclusion Criteria:

* Patients who underwent major cardiac surgeries during the hospitalization.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients' data were obtained from hospital's Clinical Data Repository (CDR), which integrates patients' baseline characteristics, laboratory results, clinical diagnosis, and treatment information during the index hospitalization. And all of the patients hospitalized from January 1,2015 to May 31,2023 in the First Affiliated Hospital of Nanjing Medical University with hs-cTnT concentrations over 14.0 ng/L were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Number of patients diagnosed with acute myocardial infarction | Within 3 days of experiencing chest pain, electrocardiogram changes, or abnormal hs-cTnT values.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roth GA, Forouzanfar MH, Moran AE, Barber R, Nguyen G, Feigin VL, Naghavi M, Mensah GA, Murray CJ. Demographic and epidemiologic drivers of global cardiovascular mortality. N Engl J Med. 2015 Apr 2;372(14):1333-41. doi: 10.1056/NEJMoa1406656. PMID 25830423
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Sandoval Y, Lewis BR, Mehta RA, Ola O, Knott JD, De Michieli L, Akula A, Lobo R, Yang EH, Gharacholou SM, Dworak M, Crockford E, Rastas N, Grube E, Karturi S, Wohlrab S, Hodge DO, Tak T, Cagin C, Gulati R, Jaffe AS. Rapid Exclusion of Acute Myocardial Injury and Infarction With a Single High-Sensitivity Cardiac Troponin T in the Emergency Department: A Multicenter United States Evaluation. Circulation. 2022 Jun 7;145(23):1708-1719. doi: 10.1161/CIRCULATIONAHA.122.059235. Epub 2022 May 10. PMID 35535607
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] Eggers KM, Hammarsten O, Aldous SJ, Cullen L, Greenslade JH, Lindahl B, Parsonage WA, Pemberton CJ, Pickering JW, Richards AM, Troughton RW, Than MP. Diagnostic and prognostic performance of the ratio between high-sensitivity cardiac troponin I and troponin T in patients with chest pain. PLoS One. 2022 Nov 1;17(11):e0276645. doi: 10.1371/journal.pone.0276645. eCollection 2022. PMID 36318533
- [Background] Nestelberger T, Boeddinghaus J, Gimenez MR, Lopez-Ayala P, Ratmann PD, Badertscher P, Wildi K, Wussler D, Koechlin L, Arslani K, Zimmermann T, Freese M, Rinderknecht T, Miro O, Martin-Sanchez FJ, Kawecki D, Geigy N, Keller D, Twerenbold R, Muller C; APACE investigators. Direct comparison of high-sensitivity cardiac troponin T and I in the early differentiation of type 1 vs. type 2 myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2022 Jan 12;11(1):62-74. doi: 10.1093/ehjacc/zuab039. PMID 34195803
- [Background] Wereski R, Kimenai DM, Taggart C, Doudesis D, Lee KK, Lowry MTH, Bularga A, Lowe DJ, Fujisawa T, Apple FS, Collinson PO, Anand A, Chapman AR, Mills NL. Cardiac Troponin Thresholds and Kinetics to Differentiate Myocardial Injury and Myocardial Infarction. Circulation. 2021 Aug 17;144(7):528-538. doi: 10.1161/CIRCULATIONAHA.121.054302. Epub 2021 Jun 25. PMID 34167318
- [Background] Collet JP, Thiele H, Barbato E, Barthelemy O, Bauersachs J, Bhatt DL, Dendale P, Dorobantu M, Edvardsen T, Folliguet T, Gale CP, Gilard M, Jobs A, Juni P, Lambrinou E, Lewis BS, Mehilli J, Meliga E, Merkely B, Mueller C, Roffi M, Rutten FH, Sibbing D, Siontis GCM; ESC Scientific Document Group. 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2021 Apr 7;42(14):1289-1367. doi: 10.1093/eurheartj/ehaa575. No abstract available. PMID 32860058
- [Background] China Society of Cardiology of Chinese Medical Association; Editorial Board of Chinese Journal of Cardiology. [Guideline for diagnosis and treatment of patients with ST-elevation myocardial infarction]. Zhonghua Xin Xue Guan Bing Za Zhi. 2010 Aug;38(8):675-90. No abstract available. Chinese. PMID 21055132